CLINICAL TRIAL: NCT01844739
Title: A Phase 1, Multiple-dose, Evaluator-blind, Randomized, Parallel Group Study Evaluating the Safety and Cutaneous Tolerability of SB204 (NVN1000 Gel) in Healthy Volunteers
Brief Title: A Phase 1 Study Evaluating Safety and Tolerability of NVN1000 Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-AC006
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Acne Vulgaris
Keywords: Propionibacterium acnes; acne
MeSH Terms: conditions — Acne Vulgaris | interventions — berdazimer sodium; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NVN1000 4% Gel (Experimental): NVN1000 4% Gel twice daily to the face for 2 weeks
  Interventions: Drug: NVN1000 4% Gel
- Vehicle Gel (Placebo Comparator): Vehicle Gel twice daily to the face for 2 weeks
  Interventions: Drug: Vehicle Gel

INTERVENTIONS:
Drug: NVN1000 4% Gel — Applied topically twice daily
  Other Names: SB204
  Arms: NVN1000 4% Gel
Drug: Vehicle Gel — Applied topically twice daily
  Other Names: Placebo
  Arms: Vehicle Gel

SUMMARY:
This is a 2 week Phase 1 study of SB204 (NVN1000 Gel) in healthy adult volunteers with elevated Propionibacterium acnes (P. acnes) counts. Subjects will apply NVN1000 4% Gel or Vehicle Gel twice daily to their face. Assessments will include cutaneous tolerability, safety, and P. acnes counts.

DETAILED DESCRIPTION:
In this single-center, vehicle gel-controlled, evaluator and subject blinded study, approximately 30 otherwise healthy adult subjects with elevated P. acnes counts will be randomized 2:1 to NVN1000 4% Gel or Vehicle Gel. The subjects will apply the test material twice daily to their face after washing. Subjects will be seen daily at the skin study center during the week and will apply their evening and weekend dose at home. Cutaneous tolerability will be assessed by the Investigator at Baseline, Week 1, and Week 2. Safety assessments include collection of adverse events, laboratory results, and clinically significant changes in physical examination. P. acnes counts will be obtained at Baseline, Week 1 and Week 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female volunteers
* If a woman of child-bearing potential, agrees to use effective method of birth control during the study and for 30 days after the final study visit
* Agree to refrain from use of antimicrobial topical products during study

Exclusion Criteria:

* Any skin disorders of acute or chronic nature including psoriasis, eczema, etc
* Female subjects who are pregnant, nursing, or planning to become pregnant
* Subjects who have used topical or systemic antibiotics, estrogens, drugs associated with methemoglobinemia, nitrate donors
* Subjects with baseline methemoglobin > 2%
* Subjects with clinically significant anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Tolerability based on the cutaneous tolerability scores | 2 weeks
  Cutaneous tolerability assessments (erythema, scaling, dryness, pruritus, burning/stinging) will be summarized with frequency counts and percentages at each score category for Week 1 and Week 2.

SECONDARY OUTCOMES:
Safety which includes reported adverse events, clinically significant changes in physical exam, and labs | 2 weeks
  Adverse events will be summarized by treatment group. Clinically significant changes in physical examination, including vital signs, over the treatment period will be reported as adverse events. Changes in laboratory results will be analyzed.

OTHER OUTCOMES:
Change in P. acnes counts | 2 weeks
  P. acnes counts will be obtained by culture at Baseline, Week 1 and Week 2/end of treatment. The change in P. acnes counts over time will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Rico, MD, Study Director — Novan, Inc.
Locations (1):
- KGL, Broomall, Pennsylvania, United States